CLINICAL TRIAL: NCT05216003
Title: Pregnancy at a Time That Is Happy and Healthy for You
Acronym: PATH4YOU
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tracey Wilkinson, Associate Professor, Department of Obstetrics & Gynecology, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1909180276
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: The study will evaluate matched-pair counties in a step-wedge design. As the intervention is implemented within a particular Indiana county, researchers will identify a matching Indiana county based on infant mortality rate. At the end of each year post-implementation, data will be compared between the intervention county and the match-paired county.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PATH4YOU County (Experimental)
  Interventions: Behavioral: PATH4YOU
- Matched-Pair Control County (No Intervention)

INTERVENTIONS:
Behavioral: PATH4YOU — PATH4YOU offers patient-center, comprehensive, contraceptive counseling; pregnancy planning; and same to next day access to birth control. This clinical care program will reduce obstacles to contraception in Indiana and enables access to healthy pregnancy planning conversations.
  Arms: PATH4YOU County

SUMMARY:
In an effort reduce maternal and infant mortality and health disparities overall, PATH4YOU (Pregnancy At a Time that's Healthy and Happy for You) will be implemented starting in Marion County, and will ultimately be a statewide comprehensive contraceptive access program that ensures that patient-centered counseling and same-day access to no (or low) cost contraception are delivered to women across the state. The goal of this project is to partner with community stakeholders to tailor and implement a patient-centered, comprehensive contraceptive access intervention, the PATH4YOU Bundle.

The health center level intervention will consist of three key principles:

1. Pregnancy Intention Screening: Provide training for health care providers and assist in health center implementation of a patient-centered pregnancy intention screening strategy within clinical settings
2. Contraception and Reproductive Health Counseling: Implement the use of a pre-visit patient-centered decision-aid for all patients presenting to a health center for reproductive health care.
3. Same-Day Access to Contraception: Provide training for health care providers and logistical assistance to health centers to implement care consistent with providing patients with their chosen method of contraception the day of patient contact.

ELIGIBILITY:
Inclusion Criteria for Clinic Level Analysis:

* women age 18-49
* presenting for care at PATH4YOU clinic site

Exclusion Criteria:

* history of hysterectomy or sterilization, or post-menopausal

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100000 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with Shared Decision Making | Within 2-4 weeks of PATH4YOU service visit
  Participant satisfaction is measured by the validated CollaboRATE scale, which is a 3 question survey. Each question is rated on a 5 point Likert scale with a response range of "every effort was made" (1) to "no effort was made" (5).
Participant Satisfaction with Same Day Contraception | Within 2-4 weeks of PATH4YOU service visit
  Participants will be asked to respond to a single question of whether they received their desired contraception on the day of the visit. Responses will be either yes or no.
Quality of family planning services | Within 2-4 weeks of PATH4YOU service visit
  Quality of family planning services will be evaluated through the validated Patient Centered Contraceptive Counseling (PCCC) Measure. The PCCC is a 4 question survey. Each question is rated on a 5 point Likert scale with responses ranging from poor (1) to excellent (5). Individual participant scores may range from 4 to 20 (with higher scores reflecting higher quality of care). A proportion of patient responses (80%) is used to determine overall quality of services. Participants will be asked to complete the PCCC one time, within 2-4 weeks after they have received care through the PATH4YOU program. Total responses will then be aggregated to determine overall quality of services upon final participant completion, approximately 3 years after project initiation.
Participant reported Pregnancy Intention | 3 months, 6 months, and 12 months
  Participants will complete the Parenting Attitudes Timing and How important (PATH) validated scale on pregnancy intention. The scale askes participants to express an opinion about having children (yes/no), to rate the importance of pregnancy on a 5 point Likert scale (from very important as a 1 to not at all important as a 5), and to estimate the timeframe in which intend to be pregnant (ranging from within 6 months to more than 5 years from now). Participants will be surveyed at 3 months, 6 months and 12 months after the PATH4YOU service visit.
Receipt of Pre-Visit Birth Control Decision Aid | Within 2-4 weeks of PATH4YOU service visit
  Participants will be asked whether they received the decision aid and whether they used it prior to the visit.
Continuation of Contraceptive Method | 3 months, 6 months, and 12 months
  Participants will be asked whether they are satisfied with, and continuation of, contraceptive method. Participants will be surveyed at 3 months, 6 months and 12 months after the PATH4YOU service visit.
Unintended pregnancy rate | 3 months, 6 months, and 12 months
  The number of unintended pregnancies within 1 year of enrollment will be assessed. Participants will be surveyed at 3 months, 6 months and 12 months after the PATH4YOU service visit.

SECONDARY OUTCOMES:
Number of women receiving PATH4YOU bundle | 3 years
  The number of participants in each county will be totaled.
Impact of demographics and reproductive characteristics | 3 years
  The sociodemographic and reproductive characteristics of participants, including participant self-reported age, race, ethnicity, gender, orientation, type of insurance, and zip code, will be evaluated to determine potential correlation with contraceptive method choice.
Contraceptive choice | 3 years
  Of the women not desiring pregnancy, the percentage of women choosing each contraceptive method will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No